CLINICAL TRIAL: NCT00062868
Title: Administration of LMP-Specific Cytotoxic T-Lymphocytes to Patients With Relapsed EBV-Positive Lymphoma (ALCI) / Previously Known as: Administration of Neomycin Resistance Gene Marked LMP2A-Specific Cytotoxic T-Lymphocytes to Patents With Relapsed EBV-Positive Lymphoma (ALASCAR)
Brief Title: LMP-specific T-cells for Patients With Relapsed EBV-positive Lymphoma
Acronym: ALCI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Helen Heslop, Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9936-ALCI-ALASCAR; ALCI (Other: Baylor College of Medicine); ALASCAR (Other: Baylor College of Medicine); NCT00070226 (obsolete NCT alias); NCT00671164 (obsolete NCT alias)
Record Dates: First submitted 2003-06-17; First posted 2003-06-18 (Estimated); Results first posted 2020-02-07 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Hodgkin Disease; Non Hodgkin Lymphoma; Lymphoepithelioma; Leiomyosarcoma
Keywords: Lymphoma; EBV-T/NK lymphoproliferative disease; Severe Chronic EBV; LMP1/2; CTL; EBV; Relapse; LMP2A
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Leiomyosarcoma; Lymphoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- LMP1/2 CTLs (ALCI - Group A) (Experimental): Patients receiving CTLs as therapy for relapsed Lymphoma/Lymphoepithelioma/leiomyosarcoma or who are at risk for relapse
  Interventions: Biological: LMP1/2 CTLs (ALCI - Group A)
- LMP1/2 CTLs (ALCI - Group B) (Experimental): Patients receiving CTLs as adjunctive therapy following autologous or syngeneic transplant.
  Interventions: Biological: LMP1/2 CTLs (ALCI - Group B)
- LMP1/2 CTLs (ALCI - Group C) (Experimental): Patients receiving CTLs following allogeneic stem cell transplant.
  Interventions: Biological: LMP1/2 CTLs (ALCI - Group C)
- LMP2A CTLs (ALASCER - Group A) (Experimental): Patients receiving CTLs as therapy for relapsed Lymphoma/Lymphoepithelioma/leiomyosarcoma or who are at risk for relapse
  Interventions: Biological: LMP2 CTLs (ALSCER - Group A)
- LMP2A CTLs (ALASCER - Group B) (Experimental): Patients receiving CTLs as adjunctive therapy following autologous or syngeneic transplant
  Interventions: Biological: LMP2 CTLs (ALSCER - Group B)
- LMP2A CTLs (ALASCER - Group C) (Experimental): Patients receiving CTLs following allogeneic stem cell transplant
  Interventions: Biological: LMP2 CTLs (ALSCER - Group C)
- LMP1/2 CTLs (ALCI - Expansion Group A) (Experimental): Patients receiving CTLs as therapy for relapsed Lymphoma/Lymphoepithelioma/leiomyosarcoma or who are at risk for relapse
  Interventions: Biological: LMP1/2 CTLs (ALCI - Expansion - Group A)
- LMP1/2 CTLs (ALCI - Expansion Group B) (Experimental): Patients receiving CTLs as adjunctive therapy following autologous or syngeneic transplant.
  Interventions: Biological: LMP1/2 CTLs (ALCI - Expansion Group B)
- LMP1/2 CTLs (ALCI - Expansion Group C) (Experimental): Patients receiving CTLs following allogeneic stem cell transplant.
  Interventions: Biological: LMP1/2 CTLs (ALCI - Expansion Group C)

INTERVENTIONS:
Biological: LMP1/2 CTLs (ALCI - Group A) — Each patient will receive 2 injections, 14 days apart, according to the following dosing schedules:
  Dose Level One
  Day 0: 2 x 10^7 cells/m2; Day 14: 2 x 10^7 cells/m2
  Dose Level Two
  Day 0: 2x10^7 cells/m2; Day 14: 1x10^8 cells/m2
  Dose Level Three
  Day 0: 1x10^8 cells/m2; Day 14: 2x10^8 cells/m2
  Arms: LMP1/2 CTLs (ALCI - Group A)
Biological: LMP1/2 CTLs (ALCI - Group B) — Each patient will receive 2 injections, 14 days apart, according to the following dosing schedules:
  Dose Level One
  Day 0: 2x10^7 cells/m2; Day 14: 2x10^7 cells/m2
  Dose Level Two
  Day 0: 2x10^7 cells/m2; Day 14: 1x10^8 cells/m2
  Dose Level Three
  Day 0: 1x10^8 cells/m2; Day 14: 2x10^8 cells/m2
  Arms: LMP1/2 CTLs (ALCI - Group B)
Biological: LMP1/2 CTLs (ALCI - Group C) — Each patient will receive 2 injections, 14 days apart, according to the following dosing schedules:
  Dose Level One
  Day 0: 2x10^7 cells/m2; Day 14: 2x10^7 cells/m2
  Dose Level Two
  Day 0: 2x10^7 cells/m2; Day 14: 1x10^8 cells/m2
  Dose Level Three
  Day 0: 1x10^8 cells/m2; Day 14: 2x10^8 cells/m2
  Arms: LMP1/2 CTLs (ALCI - Group C)
Biological: LMP2 CTLs (ALSCER - Group A) — Each patient will receive 2 injections, 14 days apart, according to the following dosing schedules:
  Dose Level One
  Day 0: 2 x 10^7 cells/m2; Day 14: 2 x 10^7 cells/m2
  Dose Level Two
  Day 0: 2x10^7 cells/m2; Day 14: 1x10^8 cells/m2
  Dose Level Three
  Day 0: 1x10^8 cells/m2; Day 14: 2x10^8 cells/m2
  Arms: LMP2A CTLs (ALASCER - Group A)
Biological: LMP2 CTLs (ALSCER - Group B) — Each patient will receive 2 injections, 14 days apart, according to the following dosing schedules:
  Dose Level One
  Day 0: 2x10^7 cells/m2; Day 14: 2x10^7 cells/m2
  Dose Level Two
  Day 0: 2x10^7 cells/m2; Day 14: 1x10^8 cells/m2
  Dose Level Three
  Day 0: 1x10^8 cells/m2; Day 14: 2x10^8 cells/m2
  Arms: LMP2A CTLs (ALASCER - Group B)
Biological: LMP2 CTLs (ALSCER - Group C) — Each patient will receive 2 injections, 14 days apart, according to the following dosing schedules:
  Dose Level One
  Day 0: 2x10^7 cells/m2; Day 14: 2x10^7 cells/m2
  Dose Level Two
  Day 0: 2x10^7 cells/m2; Day 14: 1x10^8 cells/m2
  Dose Level Three
  Day 0: 1x10^8 cells/m2; Day 14: 2x10^8 cells/m2
  Arms: LMP2A CTLs (ALASCER - Group C)
Biological: LMP1/2 CTLs (ALCI - Expansion - Group A) — Each patient will receive 2 injections, 14 days apart, according to the following dosing schedules:
  Dose Level One
  Day 0: 2 x 10^7 cells/m2; Day 14: 2 x 10^7 cells/m2
  Arms: LMP1/2 CTLs (ALCI - Expansion Group A)
Biological: LMP1/2 CTLs (ALCI - Expansion Group B) — Each patient will receive 2 injections, 14 days apart, according to the following dosing schedules:
  Dose Level One
  Day 0: 2x10^7 cells/m2; Day 14: 2x10^7 cells/m2
  Arms: LMP1/2 CTLs (ALCI - Expansion Group B)
Biological: LMP1/2 CTLs (ALCI - Expansion Group C) — Each patient will receive 2 injections, 14 days apart, according to the following dosing schedules:
  Dose Level One
  Day 0: 2x10^7 cells/m2; Day 14: 2x10^7 cells/m2
  Arms: LMP1/2 CTLs (ALCI - Expansion Group C)

SUMMARY:
This protocol is broken up into 2 portions to determine the maximum tolerated dose for treating patients with a type of lymph gland disease.

The 1st portion, called ALASCER are for people with a type of lymph gland cancer called Hodgkin or non-Hodgkin Lymphoma or Lymphoepithelioma which has returned or may return or has not gone away after treatment, including the best treatment we know for Lymphoma. While the 2nd portion (ALCI) also includes Lymphoepithelioma, severe chronic active EBV (SCAEBC), and leiomyosarcoma.

Some patients with Lymphoma show evidence of infection with the virus that causes infectious mononucleosis Epstein Barr virus (EBV) before or at the time of their diagnosis. EBV is found in the cancer cells of up to half the patients with Hodgkin's and non-Hodgkin Lymphoma, suggesting that it may play a role in causing Lymphoma. The cancer cells (in lymphoma) and some B cells (in SCAEBV) infected by EBV are able to hide from the body's immune system and escape destruction. Investigators want to see if special white blood cells, called T cells, that have been trained to kill EBV infected cells can survive in your blood and affect the tumor.

The investigators have used this sort of therapy to treat a different type of cancer that occurs after bone marrow or solid organ transplant called post transplant lymphoma. In this type of cancer the tumor cells have 9 proteins made by EBV on their surface. The investigators grew T cells in the laboratory that recognized all 9 proteins and were able to successfully prevent and treat post transplant lymphoma. However in Hodgkin disease and non-Hodgkin Lymphoma and SCAEBV, the tumor cells and B cells only express 2 EBV proteins. In a previous study we made T cells that recognized all 9 proteins and gave them to patients with Hodgkin disease. Some patients had a partial response to this therapy but no patients had a complete response. Investigators think one reason may be that many of the T cells reacted with proteins that were not on the tumor cells. In this present study we are trying to find out if we can improve this treatment by growing T cells that only recognize one of the proteins expressed on infected EBV Lymphoma cells called LMP-2a, and B cells called LMP1 and LMP2. These special T cells are called LMP specific cytotoxic T-lymphocytes (CTLs).

The purpose of the study is to find the largest safe dose of LMP specific cytotoxic T cells, to learn what the side effects are and to see whether this therapy might help patients with Hodgkin disease, non-Hodgkin Lymphoma, Lymphoepithelioma, SCAEBV or leiomyosarcoma.

DETAILED DESCRIPTION:
ALASCER (Part 1 of 2)

We will generate autologous (or syngeneic) or allogeneic LMP2A-specific cytotoxic T-cells and adoptively transfer them to patients with relapsed EBV-positive Hodgkin's or non-Hodgkins Lymphoma or Lymphoepithelioma.

To initiate the LMP-specific CTL line, PBMC will be transduced with an adenovirus vector (Ad5f35-pp65) expressing the LMP2 antigen, at a viral particle (vp) to cell ratio of 30,000:1. For blood samples from normal donors, the monocyte fraction of PBMC may be transduced and will express and present LMP2 peptide epitopes to the LMP2-specific T cell fraction of the PBMC. This step will require 20 to 40 x 106 PBMC from about 40 mL of blood.

When a stronger stimulus is required to reactivate LMP2-specific T cell precursors (i.e. from patients PBMC), then we will make dendritic cell APCs by culture of PBMC-derived monocytes with cytokines (GM-CSF, IL-4) followed by transduction with Ad5f35-LMP2 (vp:cell ratio of 30000:1) and maturation with TNF-a and PGE1. These mature, transduced dendritic cells will be used to stimulate PBMC-derived T cells. In this case, dendritic cells will be prepared from about 40 mL of blood and the T cells will be derived from 20 to 40 mL of blood

To expand the LMP2-specific T cells we will use EBV-transformed B lymphoblastoid cell lines (EBV-LCLs) transduced with Ad5f35-LMP2 (vp:LCL ratio of 100,000:1). This transduction allows the EBV-LCLs to present LMP2 peptides to the T cells. EBV-LCLs are derived from PBMC-B lymphocytes by infection with a clinical grade, laboratory strain of Epstein-Barr virus (EBV). About 5 x 106 PBMC, or 5 to 10 mLs of blood is required to generate the EBV-LCL

At the end of the CTL culture period, the frequency of LMP2 specific CTL will be determined using tetramer reagents if available.

Transduction with the Neomycin Resistance Gene (optional - based on patient preference and availability of the vector). Established CTLs will be transduced with the retroviral vectors of the LN series.

Patients will be evaluated in the clinic and 2-4 doses of CTL will be administered each two weeks apart. Patients will be monitored for clinical toxicity by the NCI Common Toxicity Criteria Scale (Version 2.0 located at http://ctep.cancer.gov). In addition, we will determine the kinetics of CTL survival by monitoring the presence of the marker gene in peripheral blood in patients who receive marked cells. We will also analyze immunological parameters including phenotype and CTL frequencies by tetramer studies in patients who have HLA types where such reagents are available. Functional analyses will be done by cytotoxicity or ELISPOT/ELISA assays. The levels of EBV DNA in peripheral blood before and following infusion will be compared. A time period of 8 weeks will constitute the time for clinical safety monitoring. If patients have had a partial response or have stable disease they will be eligible to receive up to 6 further doses of CTLs, each of which will consist of the same number as their second injection.

ALCI (Part 2 of 2)

This is the 2nd part of the ALASCER study. ALCI reflected modification in the manufacturing process to enrich the CTL product for cells recognizing the LMP1 as well as the LMP2 antigen. The change in manufacturing required to enrich for both LMP2a and LMP1 is solely to substitute ALCI's Ad5f35LMP1/2 vector for the previously used Ad5f35LMP2 vector used to transduce the antigen presenting cells used ex vivo to stimulate the T cells during the manufacturing process in our GMP laboratories.

We initially used the AD5f35LMP2 vector and now use the Ad5f35LMP1/2 vector to generate LMP-specific CTL. Our preliminary data indicates that these two vectors are identical and produce similar enrichment of LMP2 specific CTL. By using the Ad5f35LMP1/2 vector instead of the Ad5f35 vector encoding LMP2 alone, we should better enrich T cell clones recognizing both of the LMP antigens expressed by the malignant cells in Hodgkin's disease and non-Hodgkin's Lymphoma. Our analysis strategies include plans to perform comparisons between these vector types.

Like the ALASCER product, the ALCI product continued to be a CTL line specific for EBV antigens but enriched for T cells recognizing LMP1 as well as LMP2. The ALASCER product already contains some LMP1 specific T cells along with T cell specific for other EBV antigens and the only change was enrich for these cells. Therefore the ALCI Ad5f35 LMP1/2 adenoviral vector is an ancillary reagent in the manufacturing process used only to transduce antigen presenting cells used as stimulator cells and is not infused in the final product. This vector completed testing and was approved for use under ALASCER IND (#6387).

Additionally, the ALASCER protocol design was amended to allow for the addition of a separate arm to the study depending on the vector used for the manufacturing process and the data is analyzed separately

In both ALASCER & ALCI, the cells will then be thawed and injected into the patient over 10 minutes. Initially, two doses of T cells will be given two weeks apart. If after the second infusion there is a reduction in the size of the lymphoma on CT or MRI scan as assessed by a radiologist, the patient can receive up to six additional doses of the T cells if the patient wishes. This is a dose escalation study which means that for some patients the second dose may be larger than the first. All of the treatments will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or the Methodist Hospital.

The patient will be followed after the injections. They will either be seen in the clinic or will be contacted by a research nurse yearly for 5 years. To learn more about the way the T cells are working in the patient's body, an extra 20-40 mL (4-8 teaspoons) of blood will be taken before each infusion, and then 4 hours after each infusion (optional) and 3-4 days after each infusion (optional) and then weekly for 2 weeks after each infusion (total of 9 times). Two weeks after the last infusion, blood will then be taken again and then every 3 months for 1 year, then once a year for 5 years. Investigators will use this blood to see how long the T cells last and to look at the immune response to the patient's cancer.

ALCI (Expansion cohort)

Once the dose escalation safety phase of the study is completed (i.e. once at least 3 patients have been treated at dose level 3 and no treatment-related DLT has occurred), we plan to treat additional patients at dose level 1 to evaluate the immunological response in patients who receive CTL that have been generated using DC matured with the additional maturation cytokines (IL-1b and IL-6) in the presence of IL-15. We will treat an additional 30, 16, and 16 patients on Groups A, B and C, respectively.

ELIGIBILITY:
ALASCER (Part 1 of Study)

INCLUSION CRITERIA

1. Any patient, regardless of age or sex, with EBV-positive Lymphoma, or lymphoepithelioma regardless of the histological subtype or EBV (associated)-T/NK-LPD.

   In second or subsequent relapse (or first relapse or with active disease if immunosuppressive chemotherapy contraindicated or multiply relapsed patients in remission who have a high risk of relapse) OR any patient with primary disease or in first remission if immunosuppressive chemotherapy is contraindicated, e.g. patients who develop Hodgkin disease after solid organ transplantation or if the Lymphoma is a second malignancy e.g. a Richters transformation of CLL. (Group A) OR In remission or with minimal residual disease status after autologous or syngeneic SCT for Hodgkin's or non-Hodgkin's Lymphoma or lymphoepithelioma. (Group B) OR In remission or with detectable disease after allogeneic SCT. (Group C)
2. Patients with life expectancy > 6 weeks.
3. Patients with a Karnofsky/Lansky score of > 50
4. No severe intercurrent infection.
5. Donor HIV negative (if autologous product - patient must be HIV negative)
6. No evidence of GVHD > Grade II at time of enrollment.
7. If post allogeneic SCT must not have less than 50% donor chimerism in either peripheral blood or bone marrow
8. Patient, parent/guardian able to give informed consent.
9. Patients with bilirubin <3x normal, AST <5x normal, and Hgb >8.0 (see Section 7.2).
10. Patients with a creatinine <2x normal for age
11. Patients should have been off other investigational therapy for one month prior to entry in this study.

EXCLUSION CRITERIA

1. Patients with a life expectancy of <6 weeks.
2. Patients with a Karnofsky/Lansky score of < 50.
3. Patients with a severe intercurrent infection.
4. Patients with bilirubin >3x normal. AST >5x normal or abnormal prothrombin time.
5. Patients with a creatinine >2x normal for age
6. Donors who are HIV positive (Patients who are HIV positive - if autologous product)
7. Patients with GVHD Grades III-IV
8. Due to unknown effects of this therapy on a fetus, pregnant women are excluded from this research. The male partner should use a condom.

Note: Patients who would be excluded from the protocol strictly for laboratory abnormalities can be included at the investigator's discretion after approval by the CCGT Protocol Review Committee and the FDA reviewer.

ALCI and ALCI Expansion (Part 2 of Study)

INCLUSION CRITERIA:

1. Any patient, regardless of age or sex, with EBV-positive Hodgkin's or non-Hodgkin's Lymphoma, or lymphoepithelioma or leiomyosarcoma regardless of the histological subtype or EBV (associated)-T/NK-lymphoproliferative disease or Severe Chronic EBV#

   (#SCAEBV is defined as patients with high EBV viral load in plasma or PBMC (>4000 genomes per ug PBMC DNA) and/or biopsy tissue positive for EBV)

   a - In second or subsequent relapse (or first relapse or with active disease if immunosuppressive chemotherapy contraindicated or multiply relapsed patients currently in remission who have a high risk of relapse) OR with primary disease or in first or subsequent remission if immunosuppressive chemotherapy is contraindicated, e.g. patients who develop Hodgkin disease after solid organ transplantation or if the Lymphoma is a second malignancy e.g. a Richters transformation of CLL.(Group A)

   OR

   b - In remission or with minimal residual disease status after autologous or syngeneic SCT for Hodgkin's or non-Hodgkin's Lymphoma/Lymphoepithelioma/SCAEBV. (Group B)

   OR

   c - Patients in remission or with detectable disease after allogeneic SCT. (Group C)
2. Patients with life expectancy 6 weeks or greater.
3. Tumor tissue EBV positive
4. Patients with a Karnofsky/Lansky score of 50 or greater
5. Donor HIV negative (if autologous product - patient must be HIV negative)
6. If post allogeneic SCT must not have less than 50% donor chimerism in either peripheral blood or bone marrow
7. Patients with bilirubin 3x normal or less, AST 5x normal or less, and Hgb greater than 8.0
8. Patients with a creatinine 2x normal or less for age
9. Patients should have been off other investigational therapy for one month prior to entry in this study.
10. Patient, parent/guardian able to give informed consent.

EXCLUSION CRITERIA:

1. Patients with a severe intercurrent infection.
2. Donors who are HIV positive or Patients who are HIV positive if autologous product to be used
3. Patients with greater than Grade II GVHD
4. Due to unknown effects of this therapy on a fetus, pregnant women are excluded from this research. The male partner should use a condom.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2003-09 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2020-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen E Heslop, MD, Principal Investigator — Center for Cell and Gene Therapy, Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas

REFERENCES:
- [Derived] McLaughlin LP, Rouce R, Gottschalk S, Torrano V, Carrum G, Wu MF, Hoq F, Grilley B, Marcogliese AM, Hanley PJ, Gee AP, Brenner MK, Rooney CM, Heslop HE, Bollard CM. EBV/LMP-specific T cells maintain remissions of T- and B-cell EBV lymphomas after allogeneic bone marrow transplantation. Blood. 2018 Nov 29;132(22):2351-2361. doi: 10.1182/blood-2018-07-863654. Epub 2018 Sep 27. PMID 30262660
- [Derived] Bollard CM, Gottschalk S, Torrano V, Diouf O, Ku S, Hazrat Y, Carrum G, Ramos C, Fayad L, Shpall EJ, Pro B, Liu H, Wu MF, Lee D, Sheehan AM, Zu Y, Gee AP, Brenner MK, Heslop HE, Rooney CM. Sustained complete responses in patients with lymphoma receiving autologous cytotoxic T lymphocytes targeting Epstein-Barr virus latent membrane proteins. J Clin Oncol. 2014 Mar 10;32(8):798-808. doi: 10.1200/JCO.2013.51.5304. Epub 2013 Dec 16. PMID 24344220
- [Derived] Cohen JI, Jaffe ES, Dale JK, Pittaluga S, Heslop HE, Rooney CM, Gottschalk S, Bollard CM, Rao VK, Marques A, Burbelo PD, Turk SP, Fulton R, Wayne AS, Little RF, Cairo MS, El-Mallawany NK, Fowler D, Sportes C, Bishop MR, Wilson W, Straus SE. Characterization and treatment of chronic active Epstein-Barr virus disease: a 28-year experience in the United States. Blood. 2011 Jun 2;117(22):5835-49. doi: 10.1182/blood-2010-11-316745. Epub 2011 Mar 31. PMID 21454450
- [Derived] Fox CP, Haigh TA, Taylor GS, Long HM, Lee SP, Shannon-Lowe C, O'Connor S, Bollard CM, Iqbal J, Chan WC, Rickinson AB, Bell AI, Rowe M. A novel latent membrane 2 transcript expressed in Epstein-Barr virus-positive NK- and T-cell lymphoproliferative disease encodes a target for cellular immunotherapy. Blood. 2010 Nov 11;116(19):3695-704. doi: 10.1182/blood-2010-06-292268. Epub 2010 Jul 29. PMID 20671118
- [Derived] Bollard CM, Gottschalk S, Leen AM, Weiss H, Straathof KC, Carrum G, Khalil M, Wu MF, Huls MH, Chang CC, Gresik MV, Gee AP, Brenner MK, Rooney CM, Heslop HE. Complete responses of relapsed lymphoma following genetic modification of tumor-antigen presenting cells and T-lymphocyte transfer. Blood. 2007 Oct 15;110(8):2838-45. doi: 10.1182/blood-2007-05-091280. Epub 2007 Jul 3. PMID 17609424

RESULTS

PARTICIPANT FLOW:
Groups:
- LMP2A CTLs (ALASCER) - Group A DL1: Group A: Participants receiving CTLs as therapy for relapsed Lymphoma/Lymphoepithelioma/ leiomyosarcoma or who are at risk for relapse.
  Dose: Participants were administered 2 injections, 14 days apart (Day0: 2 x10^7 cells/m2, Day14: 2 x 10^7 cells/m2).
- LMP2A CTLs (ALASCER) - Group A DL2: Group A: Participants receiving CTLs as therapy for relapsed Lymphoma/Lymphoepithelioma/ leiomyosarcoma or who are at risk for relapse.
  Dose: Participants were administered 2 injections, 14 days apart (Day0: 2 x 10^7 cells/m2, Day14: 1 x 10^8 cells/m2).
- LMP2A CTLs (ALASCER) - Group A DL3: Group A: Participants receiving CTLs as therapy for relapsed Lymphoma/Lymphoepithelioma/ leiomyosarcoma or who are at risk for relapse.
  Dose: Participants were administered 2 injections, 14 days apart (Day0: 1 x 10^8 cells/m2, Day14: 2 x 10^8 cells/m2).
- LMP2A CTLs (ALASCER) - Group B DL1; LMP1/2 CTLs (ALCI) - Group B DL1; LMP1/2 CTLs (ALCI) - Group B Expansion: Group B: Participants receiving CTLs as adjunctive therapy following autologous or syngeneic transplant.
  Dose: Participants were administered 2 injections, 14 days apart (Day0: 2 x 10^7 cells/m2, Day14: 2 x 10^7 cells/m2).
- LMP2A CTLs (ALASCER) - Group B DL2; LMP1/2 CTLs (ALCI) - Group B DL2: Group B: Participants receiving CTLs as adjunctive therapy following autologous or syngeneic transplant.
  Dose: Participants were administered 2 injections, 14 days apart (Day0: 2 x 10^7 cells/m2, Day14: 1 x 10^8 cells/m2).
- LMP2A CTLs (ALASCER) - Group B DL3; LMP1/2 CTLs (ALCI) - Group B DL3: Group B: Participants receiving CTLs as adjunctive therapy following autologous or syngeneic transplant.
  Dose: Participants were administered 2 injections, 14 days apart (Day0: 1 x 10^8 cells/m2, Day14: 2 x 10^8 cells/m2).
- LMP2A CTLs (ALASCER) - Group C DL1; LMP1/2 CTLs (ALCI) - Group C DL1; LMP1/2 CTLs (ALCI) - Group C Expansion: Group C: Participants receiving CTLs following allogeneic stem cell transplant.
  Dose: Participants were administered 2 injections, 14 days apart (Day0: 2 x 10^7 cells/m2, Day14: 2 x 10^7 cells/m2).
- LMP2A CTLs (ALASCER) - Group C DL2; LMP1/2 CTLs (ALCI) - Group C DL2: Group C: Participants receiving CTLs following allogeneic stem cell transplant.
  Dose: Participants were administered 2 injections, 14 days apart (Day0: 2 x 10^7 cells/m2, Day14: 1 x 10^8 cells/m2).
- LMP2A CTLs (ALASCER) - Group C DL3; LMP1/2 CTLs (ALCI) - Group C DL3: Group C: Participants receiving CTLs following allogeneic stem cell transplant.
  Dose: Participants were administered 2 injections, 14 days apart (Day0: 1 x 10^8 cells/m2, Day14: 2 x 10^8 cells/m2).
- LMP1/2 CTLs (ALCI) - Group A DL1; LMP1/2 CTLs (ALCI) - Group A Expansion: Group A: Participants receiving CTLs as therapy for relapsed Lymphoma/ Lymphoepithelioma/ leiomyosarcoma or who are at high risk for relapse.
  Dose: Participants were administered 2 injections, 14 days apart (Day0: 2 x 10^7 cells/m2, Day14: 2 x 10^7 cells/m2).
- LMP1/2 CTLs (ALCI) - Group A DL2: Group A: Participants receiving CTLs as therapy for relapsed Lymphoma/ Lymphoepithelioma/ leiomyosarcoma or who are at high risk for relapse.
  Dose: Participants were administered 2 injections, 14 days apart (Day0: 2 x 10^7 cells/m2, Day14: 1 x 10^8 cells/m2).
- LMP1/2 CTLs (ALCI) - Group A DL3: Group A: Participants receiving CTLs as therapy for relapsed Lymphoma/ Lymphoepithelioma/ leiomyosarcoma or who are at high risk for relapse.
  Dose: Participants were administered 2 injections, 14 days apart (Day0: 1 x 10^8 cells/m2, Day14: 2 x 10^8 cells/m2).
Period: Dose Level 1
Arm/Group | LMP2A CTLs (ALASCER) - Group A DL1 | LMP2A CTLs (ALASCER) - Group A DL2 | LMP2A CTLs (ALASCER) - Group A DL3 | LMP2A CTLs (ALASCER) - Group B DL1 | LMP2A CTLs (ALASCER) - Group B DL2 | LMP2A CTLs (ALASCER) - Group B DL3 | LMP2A CTLs (ALASCER) - Group C DL1 | LMP2A CTLs (ALASCER) - Group C DL2 | LMP2A CTLs (ALASCER) - Group C DL3 | LMP1/2 CTLs (ALCI) - Group A DL1 | LMP1/2 CTLs (ALCI) - Group A DL2 | LMP1/2 CTLs (ALCI) - Group A DL3 | LMP1/2 CTLs (ALCI) - Group B DL1 | LMP1/2 CTLs (ALCI) - Group B DL2 | LMP1/2 CTLs (ALCI) - Group B DL3 | LMP1/2 CTLs (ALCI) - Group C DL1 | LMP1/2 CTLs (ALCI) - Group C DL2 | LMP1/2 CTLs (ALCI) - Group C DL3 | LMP1/2 CTLs (ALCI) - Group A Expansion | LMP1/2 CTLs (ALCI) - Group B Expansion | LMP1/2 CTLs (ALCI) - Group C Expansion
Started | 3 | 0 | 0 | 3 | 0 | 0 | 4 | 0 | 0 | 3 | 0 | 0 | 3 | 0 | 0 | 3 | 0 | 0 | 16 | 2 | 3
Completed | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 7 | 2 | 1
Not Completed | 2 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 2
Not completed — Death | 2 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Period: Dose Level 2
Arm/Group | LMP2A CTLs (ALASCER) - Group A DL1 | LMP2A CTLs (ALASCER) - Group A DL2 | LMP2A CTLs (ALASCER) - Group A DL3 | LMP2A CTLs (ALASCER) - Group B DL1 | LMP2A CTLs (ALASCER) - Group B DL2 | LMP2A CTLs (ALASCER) - Group B DL3 | LMP2A CTLs (ALASCER) - Group C DL1 | LMP2A CTLs (ALASCER) - Group C DL2 | LMP2A CTLs (ALASCER) - Group C DL3 | LMP1/2 CTLs (ALCI) - Group A DL1 | LMP1/2 CTLs (ALCI) - Group A DL2 | LMP1/2 CTLs (ALCI) - Group A DL3 | LMP1/2 CTLs (ALCI) - Group B DL1 | LMP1/2 CTLs (ALCI) - Group B DL2 | LMP1/2 CTLs (ALCI) - Group B DL3 | LMP1/2 CTLs (ALCI) - Group C DL1 | LMP1/2 CTLs (ALCI) - Group C DL2 | LMP1/2 CTLs (ALCI) - Group C DL3 | LMP1/2 CTLs (ALCI) - Group A Expansion | LMP1/2 CTLs (ALCI) - Group B Expansion | LMP1/2 CTLs (ALCI) - Group C Expansion
Started | 0 | 6 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Completed | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Dose Level 3
Arm/Group | LMP2A CTLs (ALASCER) - Group A DL1 | LMP2A CTLs (ALASCER) - Group A DL2 | LMP2A CTLs (ALASCER) - Group A DL3 | LMP2A CTLs (ALASCER) - Group B DL1 | LMP2A CTLs (ALASCER) - Group B DL2 | LMP2A CTLs (ALASCER) - Group B DL3 | LMP2A CTLs (ALASCER) - Group C DL1 | LMP2A CTLs (ALASCER) - Group C DL2 | LMP2A CTLs (ALASCER) - Group C DL3 | LMP1/2 CTLs (ALCI) - Group A DL1 | LMP1/2 CTLs (ALCI) - Group A DL2 | LMP1/2 CTLs (ALCI) - Group A DL3 | LMP1/2 CTLs (ALCI) - Group B DL1 | LMP1/2 CTLs (ALCI) - Group B DL2 | LMP1/2 CTLs (ALCI) - Group B DL3 | LMP1/2 CTLs (ALCI) - Group C DL1 | LMP1/2 CTLs (ALCI) - Group C DL2 | LMP1/2 CTLs (ALCI) - Group C DL3 | LMP1/2 CTLs (ALCI) - Group A Expansion | LMP1/2 CTLs (ALCI) - Group B Expansion | LMP1/2 CTLs (ALCI) - Group C Expansion
Started | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 3 | 0 | 0 | 4 | 0 | 0 | 0
Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The number of participants analyzed is zero if there were no participants treated in the arm/group/dose.
Groups:
- LMP1/2 CTLs (ALCI - Expansion Group A): Group A: Participants receiving CTLs as therapy for relapsed Lymphoma/ Lymphoepithelioma/ leiomyosarcoma or who are at high risk for relapse.
  Dose: Participants were administered 2 injections, 14 days apart (Day0: 2 x 10^7 cells/m2, Day14: 2 x 10^7 cells/m2).
- LMP1/2 CTLs (ALCI - Expansion Group B): Group B: Participants receiving CTLs as adjunctive therapy following autologous or syngeneic transplant.
  Dose: Participants were administered 2 injections, 14 days apart (Day0: 2 x 10^7 cells/m2, Day14: 2 x 10^7 cells/m2).
- LMP1/2 CTLs (ALCI - Expansion Group C): Group C: Participants receiving CTLs following allogeneic stem cell transplant. Dose: Participants were administered 2 injections, 14 days apart (Day0: 2 x 10^7 cells/m2, Day14: 2 x 10^7 cells/m2)
- Total: Total of all reporting groups
Arm/Group | LMP2A CTLs (ALASCER) - Group A DL1 | LMP2A CTLs (ALASCER) - Group A DL2 | LMP2A CTLs (ALASCER) - Group A DL3 | LMP2A CTLs (ALASCER) - Group B DL1 | LMP2A CTLs (ALASCER) - Group B DL2 | LMP2A CTLs (ALASCER) - Group B DL3 | LMP2A CTLs (ALASCER) - Group C DL1 | LMP2A CTLs (ALASCER) - Group C DL2 | LMP2A CTLs (ALASCER) - Group C DL3 | LMP1/2 CTLs (ALCI) - Group A DL1 | LMP1/2 CTLs (ALCI) - Group A DL2 | LMP1/2 CTLs (ALCI) - Group A DL3 | LMP1/2 CTLs (ALCI) - Group B DL1 | LMP1/2 CTLs (ALCI) - Group B DL2 | LMP1/2 CTLs (ALCI) - Group B DL3 | LMP1/2 CTLs (ALCI) - Group C DL1 | LMP1/2 CTLs (ALCI) - Group C DL2 | LMP1/2 CTLs (ALCI) - Group C DL3 | LMP1/2 CTLs (ALCI - Expansion Group A) | LMP1/2 CTLs (ALCI - Expansion Group B) | LMP1/2 CTLs (ALCI - Expansion Group C) | Total
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 3 | 0 | 4 | 0 | 0 | 3 | 4 | 5 | 3 | 3 | 3 | 3 | 3 | 4 | 16 | 2 | 3 | 74
Age, Continuous [Median (Full Range); unit: years] | 39 [32 to 49] | 53 [19 to 69] | 13 [7 to 15] | 57 [7 to 66] | 25 [17 to 52] |  | 54 [26 to 59] |  |  | 46 [21 to 69] | 54 [18 to 79] | 55 [28 to 62] | 23 [18 to 34] | 18 [14 to 38] | 43 [24 to 64] | 13 [10 to 43] | 30 [14 to 33] | 17.5 [6 to 51] | 45 [6 to 78] | 39 [31 to 47] | 16 [12 to 23] | 33.5 [6 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 2 | 1 |  | 1 |  |  | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 2 | 7 | 0 | 2 | 27
  Male | 1 | 4 | 2 | 1 | 2 |  | 3 |  |  | 2 | 4 | 3 | 3 | 3 | 2 | 2 | 1 | 2 | 9 | 2 | 1 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 0 | 0 |  | 0 |  |  | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 2 | 0 | 4 | 0 | 0 | 14
  Not Hispanic or Latino | 3 | 6 | 1 | 3 | 3 |  | 4 |  |  | 3 | 3 | 4 | 3 | 2 | 2 | 1 | 1 | 4 | 12 | 1 | 3 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 |  | 0 |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian | 0 | 0 | 0 | 0 | 0 |  | 0 |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Asian | 0 | 0 | 0 | 1 | 0 |  | 0 |  |  | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5
  Black or African American | 0 | 2 | 0 | 0 | 0 |  | 0 |  |  | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 6
  White | 3 | 4 | 3 | 2 | 3 |  | 4 |  |  | 1 | 3 | 4 | 3 | 3 | 1 | 2 | 2 | 4 | 12 | 1 | 2 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 |  | 0 |  |  | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT) Rate by the NCI Common Toxicity Criteria (CTCAE) v2.0 and the Method of Przepiorka et al (Protocol Appendix I)
Description: Dose limiting toxicity (DLT) rate is the proportion of participants with DLT. DLT will be defined as any toxicity that is irreversible, life threatening or Grade 3-4 considered to be primarily related to the LMP-specific cytotoxic T-lymphocytes (CTL) injection or development of Grade III-IV Graft versus host disease (GVHD). Toxicity will be evaluated according to the CTCAE Version 2.0. GVHD will be graded by the method of Przepiorka et al (protocol Appendix I).
Time Frame: 6 weeks post second CLT infusion
Population: Data is reported for all DLT evaluable participants who received CTL infusions and either completed the DLT assessment period or dropped off the study early due to DLT. One participant in the LMP1/2 CTLs (ALCI) - Group A Expansion was enrolled to this arm/group twice. DLT assessment data from the first enrollment is reported for this participant.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | LMP2A CTLs (ALASCER) - Group A DL1 | LMP2A CTLs (ALASCER) - Group A DL2 | LMP2A CTLs (ALASCER) - Group A DL3 | LMP2A CTLs (ALASCER) - Group B DL1 | LMP2A CTLs (ALASCER) - Group B DL2 | LMP2A CTLs (ALASCER) - Group B DL3 | LMP2A CTLs (ALASCER) - Group C DL1 | LMP2A CTLs (ALASCER) - Group C DL2 | LMP2A CTLs (ALASCER) - Group C DL3 | LMP1/2 CTLs (ALCI) - Group A DL1 | LMP1/2 CTLs (ALCI) - Group A DL2 | LMP1/2 CTLs (ALCI) - Group A DL3 | LMP1/2 CTLs (ALCI) - Group B DL1 | LMP1/2 CTLs (ALCI) - Group B DL2 | LMP1/2 CTLs (ALCI) - Group B DL3 | LMP1/2 CTLs (ALCI) - Group C DL1 | LMP1/2 CTLs (ALCI) - Group C DL2 | LMP1/2 CTLs (ALCI) - Group C DL3 | LMP1/2 CTLs (ALCI) - Group A Expansion | LMP1/2 CTLs (ALCI) - Group B Expansion | LMP1/2 CTLs (ALCI) - Group C Expansion
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 3 | 0 | 3 | 0 | 0 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 15 | 2 | 2
proportion of participants | 0 [0 to 0.708] | 0 [0 to 0.459] | 0 [0 to 0.708] | 0 [0 to 0.708] | 0 [0 to 0.708] |  | 0 [0 to 0.708] |  |  | 0 [0 to 0.708] | 0 [0 to 0.708] | 0 [0 to 0.602] | 0 [0 to 0.708] | 0 [0 to 0.708] | 0 [0 to 0.708] | 0 [0 to 0.708] | 0 [0 to 0.708] | 0 [0 to 0.602] | 0 [0 to 0.218] | 0 [0 to 0.842] | 0 [0 to 0.842]

2. Secondary Outcome: Response Rate According to the Harmonization Project (Protocol 8.5.1) or RECIST Criteria.
Description: Response rate is defined as the proportion of participants with best overall response of complete response (CR) or partial response (PR) . All patients who receive the first infusion will be evaluable for response.
  In patients with detectable tumors and/or lymphadenopathy - response and progression will be evaluated using PET based imaging studies (whenever possible) based on the Harmonization Project (protocol 8.5.1). All available non-PET imaging studies will be evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee.
Time Frame: Up to 4 months after the last infusion
Population: Data is reported for all participants who has received at least one infusion and has available response assessment data. One participant in LMP1/2 CTLs (ALCI) - Group A Expansion is excluded because of no available response data and one was enrolled to this arm/group twice that response assessment data from the first enrollment is reported.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | LMP2A CTLs (ALASCER) - Group A DL1 | LMP2A CTLs (ALASCER) - Group A DL2 | LMP2A CTLs (ALASCER) - Group A DL3 | LMP2A CTLs (ALASCER) - Group B DL1 | LMP2A CTLs (ALASCER) - Group B DL2 | LMP2A CTLs (ALASCER) - Group B DL3 | LMP2A CTLs (ALASCER) - Group C DL1 | LMP2A CTLs (ALASCER) - Group C DL2 | LMP2A CTLs (ALASCER) - Group C DL3 | LMP1/2 CTLs (ALCI) - Group A DL1 | LMP1/2 CTLs (ALCI) - Group A DL2 | LMP1/2 CTLs (ALCI) - Group A DL3 | LMP1/2 CTLs (ALCI) - Group B DL1 | LMP1/2 CTLs (ALCI) - Group B DL2 | LMP1/2 CTLs (ALCI) - Group B DL3 | LMP1/2 CTLs (ALCI) - Group C DL1 | LMP1/2 CTLs (ALCI) - Group C DL2 | LMP1/2 CTLs (ALCI) - Group C DL3 | LMP1/2 CTLs (ALCI) - Group A Expansion | LMP1/2 CTLs (ALCI) - Group B Expansion | LMP1/2 CTLs (ALCI) - Group C Expansion
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 3 | 0 | 4 | 0 | 0 | 3 | 4 | 5 | 3 | 3 | 3 | 3 | 3 | 4 | 15 | 2 | 3
proportion of participants | 0.667 [0.094 to 0.992] | 0.833 [0.359 to 0.996] | 0.667 [0.094 to 0.992] | 0.333 [0.008 to 0.906] | 0.667 [0.094 to 0.992] |  | 0.75 [0.194 to 0.994] |  |  | 1 [0.292 to 1] | 0.75 [0.194 to 0.994] | 0.6 [0.147 to 0.947] | 1 [0.292 to 1] | 1 [0.292 to 1] | 1 [0.292 to 1] | 1 [0.292 to 1] | 0.667 [0.094 to 0.992] | 1 [0.398 to 1] | 0.733 [0.449 to 0.922] | 0.5 [0.013 to 0.987] | 0.333 [0.008 to 0.906]

3. Secondary Outcome: Grade III-IV Toxicity Rate in Participants Receiving an Extended Dosage Regimen According to the NCI Common Toxicity Criteria (CTCAE) Version 2.0 and the Method of Przepiorka et. al. (Protocol Appendix I).
Description: Grade III-IV toxicity rate is defined as the proportion of participants who receive an extended dose regimen and developed Grade III-IV toxicity attributable to the CTL infusions at any time during the extended dosing regimen. Toxicity will be evaluated according to the CTCAE Version 2.0. GVHD will be graded by the method of Przepiorka et al (protocol Appendix I).
Time Frame: 6 weeks after the final injection
Population: Data is reported for participants who have received an extended dosage regimen.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | LMP2A CTLs (ALASCER) - Group A DL1 | LMP2A CTLs (ALASCER) - Group A DL2 | LMP2A CTLs (ALASCER) - Group A DL3 | LMP2A CTLs (ALASCER) - Group B DL1 | LMP2A CTLs (ALASCER) - Group B DL2 | LMP2A CTLs (ALASCER) - Group B DL3 | LMP2A CTLs (ALASCER) - Group C DL1 | LMP2A CTLs (ALASCER) - Group C DL2 | LMP2A CTLs (ALASCER) - Group C DL3 | LMP1/2 CTLs (ALCI) - Group A DL1 | LMP1/2 CTLs (ALCI) - Group A DL2 | LMP1/2 CTLs (ALCI) - Group A DL3 | LMP1/2 CTLs (ALCI) - Group B DL1 | LMP1/2 CTLs (ALCI) - Group B DL2 | LMP1/2 CTLs (ALCI) - Group B DL3 | LMP1/2 CTLs (ALCI) - Group C DL1 | LMP1/2 CTLs (ALCI) - Group C DL2 | LMP1/2 CTLs (ALCI) - Group C DL3 | LMP1/2 CTLs (ALCI) - Group A Expansion | LMP1/2 CTLs (ALCI) - Group B Expansion | LMP1/2 CTLs (ALCI) - Group C Expansion
Number analyzed (Participants) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
proportion of participants | 0 [0 to 0.842] | 0 [0 to 0.975] | 0 [0 to 0.975] |  |  |  |  |  |  | 0 [0 to 0.975] |  | 0 [0 to 0.975] |  |  |  |  |  |  | 0 [0 to 0.975] |  |

ADVERSE EVENTS:
Time Frame: Data on adverse experiences/toxicities regardless of seriousness were collected for documentation purposes only for 6 weeks after the last dosing of the study drug/biologic.
Description: Zeros in the number of participants at risk for Other/Serious Adverse Events and the number of participants at risk for All-Cause Mortality are due to no participants treated at those arms/groups.
  One participant in the LMP1/2 CTLs (ALCI) - Group A Expansion was enrolled to this arm/group twice. All adverse event data is included for this participant regardless of enrollment.
Arm/Group | LMP2A CTLs (ALASCER) - Group A DL1 | LMP2A CTLs (ALASCER) - Group A DL2 | LMP2A CTLs (ALASCER) - Group A DL3 | LMP2A CTLs (ALASCER) - Group B DL1 | LMP2A CTLs (ALASCER) - Group B DL2 | LMP2A CTLs (ALASCER) - Group B DL3 | LMP2A CTLs (ALASCER) - Group C DL1 | LMP2A CTLs (ALASCER) - Group C DL2 | LMP2A CTLs (ALASCER) - Group C DL3 | LMP1/2 CTLs (ALCI) - Group A DL1 | LMP1/2 CTLs (ALCI) - Group A DL2 | LMP1/2 CTLs (ALCI) - Group A DL3 | LMP1/2 CTLs (ALCI) - Group B DL1 | LMP1/2 CTLs (ALCI) - Group B DL2 | LMP1/2 CTLs (ALCI) - Group B DL3 | LMP1/2 CTLs (ALCI) - Group C DL1 | LMP1/2 CTLs (ALCI) - Group C DL2 | LMP1/2 CTLs (ALCI) - Group C DL3 | LMP1/2 CTLs (ALCI) - Group A Expansion | LMP1/2 CTLs (ALCI) - Group B Expansion | LMP1/2 CTLs (ALCI) - Group C Expansion
All-Cause Mortality (participants affected / at risk) | 2/3 | 3/6 | 0/3 | 2/3 | 2/3 | 0/0 | 3/4 | 0/0 | 0/0 | 0/3 | 1/4 | 1/5 | 0/3 | 0/3 | 0/3 | 0/3 | 2/3 | 1/4 | 7/16 | 0/2 | 1/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/6 | 0/3 | 1/3 | 0/3 | 0/0 | 1/4 | 0/0 | 0/0 | 0/3 | 1/4 | 1/5 | 0/3 | 1/3 | 0/3 | 1/3 | 0/3 | 1/4 | 3/16 | 0/2 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 3/3 | 3/3 | 3/3 | 0/0 | 4/4 | 0/0 | 0/0 | 3/3 | 4/4 | 5/5 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 4/4 | 16/16 | 2/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LMP2A CTLs (ALASCER) - Group A DL1 (N=3) | LMP2A CTLs (ALASCER) - Group A DL2 (N=6) | LMP2A CTLs (ALASCER) - Group A DL3 (N=3) | LMP2A CTLs (ALASCER) - Group B DL1 (N=3) | LMP2A CTLs (ALASCER) - Group B DL2 (N=3) | LMP2A CTLs (ALASCER) - Group B DL3 (N=0) | LMP2A CTLs (ALASCER) - Group C DL1 (N=4) | LMP2A CTLs (ALASCER) - Group C DL2 (N=0) | LMP2A CTLs (ALASCER) - Group C DL3 (N=0) | LMP1/2 CTLs (ALCI) - Group A DL1 (N=3) | LMP1/2 CTLs (ALCI) - Group A DL2 (N=4) | LMP1/2 CTLs (ALCI) - Group A DL3 (N=5) | LMP1/2 CTLs (ALCI) - Group B DL1 (N=3) | LMP1/2 CTLs (ALCI) - Group B DL2 (N=3) | LMP1/2 CTLs (ALCI) - Group B DL3 (N=3) | LMP1/2 CTLs (ALCI) - Group C DL1 (N=3) | LMP1/2 CTLs (ALCI) - Group C DL2 (N=3) | LMP1/2 CTLs (ALCI) - Group C DL3 (N=4) | LMP1/2 CTLs (ALCI) - Group A Expansion (N=16) | LMP1/2 CTLs (ALCI) - Group B Expansion (N=2) | LMP1/2 CTLs (ALCI) - Group C Expansion (N=3)
Nodal/junctional arrhythmia/dysrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac-ischemia/infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound-Infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bilirubin (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 10e (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection without neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness/lightheadedness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy - Motor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary-Other:pulmonaryembolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Secondary Malignancy-Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SecondaryMalignancy-Other:PERIPHERALPRIMITIVENEUROECTODERMALTUMOR/ EWINGSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SecondaryMalignancy-Other:SpindleCellSarcoma-periaortic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SecondaryMalignancy-Other:Squamouscellcarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LMP2A CTLs (ALASCER) - Group A DL1 (N=3) | LMP2A CTLs (ALASCER) - Group A DL2 (N=6) | LMP2A CTLs (ALASCER) - Group A DL3 (N=3) | LMP2A CTLs (ALASCER) - Group B DL1 (N=3) | LMP2A CTLs (ALASCER) - Group B DL2 (N=3) | LMP2A CTLs (ALASCER) - Group B DL3 (N=0) | LMP2A CTLs (ALASCER) - Group C DL1 (N=4) | LMP2A CTLs (ALASCER) - Group C DL2 (N=0) | LMP2A CTLs (ALASCER) - Group C DL3 (N=0) | LMP1/2 CTLs (ALCI) - Group A DL1 (N=3) | LMP1/2 CTLs (ALCI) - Group A DL2 (N=4) | LMP1/2 CTLs (ALCI) - Group A DL3 (N=5) | LMP1/2 CTLs (ALCI) - Group B DL1 (N=3) | LMP1/2 CTLs (ALCI) - Group B DL2 (N=3) | LMP1/2 CTLs (ALCI) - Group B DL3 (N=3) | LMP1/2 CTLs (ALCI) - Group C DL1 (N=3) | LMP1/2 CTLs (ALCI) - Group C DL2 (N=3) | LMP1/2 CTLs (ALCI) - Group C DL3 (N=4) | LMP1/2 CTLs (ALCI) - Group A Expansion (N=16) | LMP1/2 CTLs (ALCI) - Group B Expansion (N=2) | LMP1/2 CTLs (ALCI) - Group C Expansion (N=3)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Allergy/Immunology-Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy/Immunology-Other:Sorethroat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy/Immunology-Other:excessmucus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy/Immunology-Other:lymphnodeswelling (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy/Immunology-Other:moresignificanthistaminereaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Auditory/Hearing-Other (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin-Hgb (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 3 (3) | 1 (8) | 2 (6) | 1 (2) | 2 (4) | 1 (2) | 1 (1) | 2 (12) | 2 (8) | 7 (16) | 0 (0) | 2 (4)
Leukocytes (total WBC) (Investigations) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (5) | 3 (4) | 3 (8) | 2 (14) | 2 (3) | 3 (8) | 2 (23) | 3 (23) | 13 (26) | 2 (2) | 2 (4)
Leukopenia (total WBC) (Investigations) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Investigations) | 0 (0) | 5 (15) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 1 (2) | 2 (5) | 4 (7) | 3 (6) | 1 (10) | 2 (5) | 2 (3) | 3 (9) | 2 (18) | 10 (28) | 1 (1) | 1 (3)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2 (6) | 4 (5) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 2 (8) | 0 (0) | 0 (0) | 1 (2) | 1 (9) | 3 (3) | 2 (5) | 2 (17) | 1 (1) | 3 (8) | 2 (24) | 3 (24) | 9 (17) | 0 (0) | 2 (2)
Platelets (Investigations) | 2 (5) | 2 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (12) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 1 (8) | 3 (9) | 6 (13) | 0 (0) | 0 (0)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Transfusion; Platelets (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion; pRBC's (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrinogen (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Partial thromboplastin time (PTT) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prothrombin time (PT) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constitutional Symptoms-Other (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 0 (0) | 3 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (7) | 0 (0) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Fever-absence of Neutropenia (General disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rigors, chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rigors/Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sweating (Diaphoresis) (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sweating (diaphoresis) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death not associated with CTCAE term - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (absence of thrombocytopenia grade 3/4) (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (in absence of grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin-Other:Face&neckpimples (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dermatology/Skin-Other:SpongioticDermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin-Other:pimples (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 2 (3) | 0 (0) | 0 (0)
Wound-Infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot Flashes/Flushes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (without colostomy) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia/Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal-Other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal-Other:erythemaofpharynx (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disturbance (dysgeusia) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage/Bleeding w/gr 3/4 Thrombocytopenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae/Purpura(hemorrhage/bleeding skin/mucosa) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bilirubin (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Hepatic-Other:Hypoproteinemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 4 (4) | 0 (0) | 1 (2)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 2 (6) | 2 (2) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 3 (11) | 2 (4) | 5 (8) | 1 (2) | 2 (3)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alkaline Phosphatase (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic-Other (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SGOT(AST) (serum glutamic oxal. Transaminase) (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (3) | 1 (1) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SGPT(ALT) (seurm glutamic pyruric trans.) (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 10e (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Infection without Neutropenia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection without neutropenia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (6) | 11 (14) | 0 (0) | 3 (6)
Lymphatics-Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphatics-Other:cervicaladenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amylase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bicarbonate (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (4) | 4 (5) | 2 (2) | 1 (2) | 1 (1) | 2 (4) | 2 (3) | 2 (3) | 2 (10) | 2 (2) | 0 (0) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (4) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (10) | 2 (11) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 3 (7) | 0 (0) | 2 (12) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (3) | 2 (4) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (11) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 4 (5) | 2 (3) | 1 (1) | 1 (2) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (2) | 2 (6) | 3 (5) | 1 (1) | 2 (3) | 0 (0) | 1 (3) | 2 (12) | 2 (11) | 4 (8) | 1 (1) | 2 (2)
Hypomagnesmia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (6) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (3) | 0 (0) | 2 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic/Laboratory-Other (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic/Laboratory-Other:Hyperchloremia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic/Laboratory-Other:Hypochloremia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskelatal-Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dizziness/Lightheadedness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness/lightheadedness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood alteration-anxiety, agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurology-Other:Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy - motor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy-Sensory (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular-Visual Other (Eye disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular/Visual-Other:Periorbitalerythemaandswelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular/Visual-Other:Visionhaziness (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tearing (watery eyes) (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain or Cramping (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain or cramping (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (non-cardiac, non-pleuritic) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (non-cardiac and non-pleuritic) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Neuropathic Pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain-Other (General disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain-Other:Ankle,backandknee (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain-Other:Legpain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain-Other:Oralpain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain-Other:SORETHROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain-Other:bodyaches (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain-Other:generalizedaches&pains (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain-Other:lefthandpain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain-Other:leftshoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain-Other:upperrightarm (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (onset or exacerbation of tumor pain due to treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary-Other:Reactiveairwaydisease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary-Other:SORETHROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary-Other:Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Voice changes/stridor/larynx (e.g., hoarseness, loss of voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary-Other:RespiratoryFailure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary-Other:sorethroat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Voice changes/stridor/larynx (e.g., hoarseness, loss of voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 2 (4) | 2 (5) | 0 (0) | 0 (0)
Dysuria (painful urination) (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal/Genitourinary-Other (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal/Genitourinary-Other:BUN (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Frequency/Urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SecondaryMalignancy-Other:Highgradesarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SecondaryMalignancy-Other:MyelodysplasticSyndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SecondaryMalignancy-Other:squamouscellcarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes